CLINICAL TRIAL: NCT02941055
Title: ADIRA (Anti-inflammatory Diet In Rheumatoid Arthritis)
Acronym: ADIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ADIRA2016
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Diet; Inflammation; Metabolomics
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber diet (Experimental): 50% of daily intake, 5 days a week, a diet rich in fiber, fish and probiotics will be provided to study subjects
  Interventions: Other: Fiber diet
- Protein diet (Active Comparator): 50% of daily intake, 5 days a week, a diet rich in protein, red meat and saturated fat will be provided to study subjects
  Interventions: Other: Protein diet

INTERVENTIONS:
Other: Fiber diet — Foods will be delivered with a home delivery chain once a week for 10 wks of each diet
  Arms: Fiber diet
Other: Protein diet — Foods will be delivered with a home delivery chain once a week for 10 wks of each diet
  Arms: Protein diet

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that affects 0.5-1% of the population, and where many patients in spite of modern pharmacological treatment fail to reach remission. The main goal of the randomized cross-over trial ADIRA (Anti-inflammatory Diet In Rheumatoid Arthritis) is to test the hypothesis that a diet intervention will decrease disease activity and improve quality of life in patients with established RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that affects 0.5-1% of the population, and where many patients in spite of modern pharmacological treatment fail to reach remission. This affects physical as well as mental wellbeing and leads to severely reduced quality of life and reduced work capacity, thus yielding high individual as well as societal costs. To optimize treatment, alternatives such as diet should be evaluated as complement to pharmacological treatment. The main goal of the randomized cross-over trial ADIRA (Anti-inflammatory Diet In Rheumatoid Arthritis) is to test the hypothesis that a diet intervention will decrease disease activity and costs and improve quality of life in patients with established RA. In total, 60 RA patients with moderate disease activity will be randomized to receive initially either a portfolio diet based on several food items with suggested anti-inflammatory effects or a control diet (western type), during 2 x 10 wks with a 3 months wash-out between diets. Both groups continue with regular pharmacological treatment. Known food biomarkers will be analyzed to measure intervention compliance. Impact on disease activity (measured by DAS28, a composite score which predicts disability and progression of RA) and quality of life is evaluated after each diet regimen. Metabolomics will be used to evaluate the potential to predict responders to dietary treatment. ADIRA will provide evidence whether dietary treatment of RA leads to more patients reaching remission and improved quality of life and work capacity as well as reduce individual and societal costs. Scientific evidence exists for anti-inflammatory effect by single foods on RA, but no study exists where these foods have been combined to obtain maximum effect and thus have the potential to offer a substantial improvement in patient life quality. Such evidence has been asked for by RA patents as well as by treating physicians.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with established RA, disease duration >2 years, disease activity DAS28 >= 2.6 and a disease that is clinically stable and under adequate control and medication, will be invited to participate.

Exclusion Criteria:

* Other life threatening diseases, pregnancy, lactation, food intolerance or allergy to food included in the trial, ability to understand information in Swedish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Difference in disease activity score DAS28 (ie a composite score including tender and swollen joints count, ESR or CRP, VAS scale global health) between the two diet interventions, within each person | 10 weeks of each diet
  Measured clinically

SECONDARY OUTCOMES:
Difference in SF-36 between the two diet interventions, within each person | 10 weeks on each diet
  Measured by validated instruments
Difference and changes in metabolites between the two diet interventions, within each person | 10 weeks on each diet
  Metabolomics with NMR and MS analyses of serum and urine samples
Differences in inflammatory markers between the two diet interventions, within each person | 10 weeks on each diet
  hs-CRP, cytokines in blood
Difference in EQ5D between the two diet interventions, within each person | 10 weeks on each diet
  Measured by validated instruments
Difference in HAQ between the two diet interventions, within each person | 10 weeks on each diet
  Measured by validated instruments

OTHER OUTCOMES:
Cost effectiveness of study intervention by Health-related quality of life | 10 weeks on each diet
  Health-related quality of life
Cost effectiveness of study intervention by QALYs | 10 weeks on each diet
  Quality-adjusted life years (QALYs)
Changes in blood lipids between the two diet interventions, within each person | 10 weeks on each diet
  TAG, LDL, HDL etc
Effects of genetic polymorphisms in dietary response | 10 weeks on each diet
  Genetic analyses

CONTACTS AND LOCATIONS:
Overall Officials: Anna Winkvist, PhD, Principal Investigator — Göteborg University
Locations (1):
- The University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Not approved by the Ethical Review board

REFERENCES:
- [Background] Winkvist A, Barebring L, Gjertsson I, Ellegard L, Lindqvist HM. A randomized controlled cross-over trial investigating the effect of anti-inflammatory diet on disease activity and quality of life in rheumatoid arthritis: the Anti-inflammatory Diet In Rheumatoid Arthritis (ADIRA) study protocol. Nutr J. 2018 Apr 20;17(1):44. doi: 10.1186/s12937-018-0354-x. PMID 29678183
- [Result] Barebring L, Winkvist A, Gjertsson I, Lindqvist HM. Poor Dietary Quality Is Associated with Increased Inflammation in Swedish Patients with Rheumatoid Arthritis. Nutrients. 2018 Oct 18;10(10):1535. doi: 10.3390/nu10101535. PMID 30340316
- [Derived] Wadell AT, Barebring L, Hulander E, Gjertsson I, Landberg R, Lindqvist H, Winkvist A. Dietary biomarkers and food records indicate compliance to study diets in the ADIRA (Anti-inflammatory Diet In Rheumatoid Arthritis) trial. Front Nutr. 2023 Jun 22;10:1209787. doi: 10.3389/fnut.2023.1209787. eCollection 2023. PMID 37426179
- [Derived] Turesson Wadell A, Barebring L, Hulander E, Gjertsson I, Lindqvist HM, Winkvist A. Inadequate Dietary Nutrient Intake in Patients With Rheumatoid Arthritis in Southwestern Sweden: A Cross-Sectional Study. Front Nutr. 2022 Jun 21;9:915064. doi: 10.3389/fnut.2022.915064. eCollection 2022. PMID 35799579
- [Derived] Hulander E, Barebring L, Turesson Wadell A, Gjertsson I, Calder PC, Winkvist A, Lindqvist HM. Diet intervention improves cardiovascular profile in patients with rheumatoid arthritis: results from the randomized controlled cross-over trial ADIRA. Nutr J. 2021 Jan 23;20(1):9. doi: 10.1186/s12937-021-00663-y. PMID 33485336
- [Derived] Vadell AKE, Barebring L, Hulander E, Gjertsson I, Lindqvist HM, Winkvist A. Anti-inflammatory Diet In Rheumatoid Arthritis (ADIRA)-a randomized, controlled crossover trial indicating effects on disease activity. Am J Clin Nutr. 2020 Jun 1;111(6):1203-1213. doi: 10.1093/ajcn/nqaa019. PMID 32055820